CLINICAL TRIAL: NCT01671449
Title: Phase III Trial of S-1 and Cisplatin (3 Weekly) Versus S-1 and Oxaliplatin Combination Chemotherapy for First Line Treatment of Advanced Gastric Cancer
Brief Title: S-1 and Cisplatin (3 Weekly) Versus S-1 and Oxaliplatin Combination Chemotherapy for Advanced Gastric Cancer
Acronym: SOPP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Min-Hee Ryu (Other)
Responsible Party: Sponsor-Investigator, Min-Hee Ryu, Asan Medical Center, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC-ONCGI-1202
Record Dates: First submitted 2012-08-17; First posted 2012-08-23 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; S-1; Cisplatin; Oxaliplatin
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); titanium silicide; Cisplatin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-1 plus Cisplatin (Active Comparator): * S-1: 40 mg/m2, twice daily, p.o., day 1-14 (see Table 6 for dose calculation of S-1 according to body surface area)
    : If S-1 is started on the evening of day 1, last dose of S-1 will be administered at the morning of day 15.
  * Cisplatin: 60 mg/ m2/day, i.v., day 1
  * Every 3 weeks
  Interventions: Drug: S-1; Drug: Cisplatin
- S-1 plus Oxaliplatin (Experimental): * S-1: 40 mg/m2, twice daily, p.o., day 1-14 (see Table 6 for dose calculation of S-1 according to body surface area)
    : If S-1 is started on the evening of day 1, last dose of S-1 will be administered at the morning of day 15.
  * Oxaliplatin: 130 mg/ m2/day, i.v., day 1
  * Every 3 weeks
  Interventions: Drug: S-1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: S-1 — S-1 : 40 mg/m2, twice daily, Day 1-14
  Other Names: TS-1
Drug: Cisplatin — 60 mg/m2/day Day 1
  Arms: S-1 plus Cisplatin
Drug: Oxaliplatin — 130 mg/m2/day Day 1
  Other Names: Pleoxin
  Arms: S-1 plus Oxaliplatin

SUMMARY:
A multicenter, randomized, open-label, phase III trial of S-1 plus cisplatin (3 weekly) versus S-1 plus oxaliplatin chemotherapy for the first-line treatment of advanced gastric cancer

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent before the enrollment
2. Age ≥18 years old
3. Histologically/cytologically confirmed recurrent or metastatic gastric or esophagogastric junctional adenocarcinoma
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
5. Patients able to swallow food and drugs
6. At least one measurable or evaluable lesion according to RECIST criteria version 1.1
7. Adequate bone, hepatic, and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to first administration of study drugs

   * Absolute neutrophil count (ANC) ≥ 1,500/ uL, platelet ≥ 100,000/ uL, haemoglobin (Hb) ≥ 9.0 g/dl,
   * Serum creatinine ≤ 1.5 mg/dL (If serum creatinine is greater than 1.5 mg/dL, creatinine clearance [Ccr] should be 60 mL/min or greater. Ccr is calculated by Cockcroft-Gault formula or 24hr urine collection)
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN), AST/ALT levels ≤ 3.0 x ULN (AST/ALT levels ≤ 5.0 x ULN for patients with liver involvement of their cancer)
8. In patients who received adjuvant or neoadjuvant chemotherapy, completion of systemic chemotherapy 6 months before the study enrollment, and no previous administration of platinum derivatives
9. Estimated life expectancy of more than 3 months

Exclusion Criteria:

1. Other histologic types than adenocarcinoma
2. Recurrence within 24 weeks following completion of adjuvant chemotherapy
3. R1 gastrectomy (i.e., microscopic residual disease)
4. History of another malignancy within the last five years from the day of written informed consent except cured basal cell carcinoma of skin and cured carcinoma in situ of uterine cervix
5. Radiotherapy within 4 weeks after randomization
6. History of significant neurologic or psychiatric disorders, and presence or history of CNS metastasis
7. Major surgery within 4 weeks before study entry, or insufficient recovery from major surgery (except the patients who received only open and closure or biopsy)
8. Other serious illness or medical conditions as follows;

   * Any following conditions occurred within 6 months before study entry: myocardial infarction, severe/unstable angina, bypass surgery for coronary artery/peripheral artery, congestive heart failure (NYHA class III or IV), cerebral infarction or transient ischemic attack
   * Conduction abnormality such as 2nd degree or greater AV block or severe arrhythmia that requires medical treatments (right bundle branch block (RBBB) is eligible, but left bundle branch block (LBBB) is not.)
   * Uncontrolled hypertension
   * Liver cirrhosis (Child Pugh Class B or greater)
   * Interstitial pneumonia, pulmonary fibrosis
   * Active viral hepatitis B
   * Uncontrolled diabetes mellitus
   * Uncontrolled ascites or pleural effusion
   * Uncontrolled active infection or sepsis
9. Administration of medications which may have potentially pharmacokinetic interaction with S-1, cisplatin, and oxaliplatin

   * Flucytosine, a fluorinated pyrimidine antifungal agent
   * Anti-viral agents, such as sorivudine, and brivudine, or chemical similar drugs
   * Warfarin (except, low dose warfarin for the purpose of prophylaxis), phenprocoumon
   * Phenytoin
   * Allopurinol
10. Participation to other clinical trials or administration of other investigational drugs within 30 days before the randomisation
11. Pregnant or lactating women
12. Women or men of child bearing potential not employing adequate contraception during study treatments or until the 3 months after the end of study treatments
13. Ineligible for the study at the discretion of investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  The primary endpoint of this study is progression-free survival. This is defined as the time from randomization to disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall survival | From date of randomization to death from any cause, assessed up to 3 years
  Overall survival is defined as the time from randomization to death due to any cause.
Response rate | Every 6 weeks
  Response assessment will be performed according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 every 2 cycles (6 weeks) of treatment.
Quality of life | Every 6 weeks
  Quality of life of patient will be evaluated using EUROQOL(EQ-5D). Evaluation of quality of life will be performed every 2 cycles (6 weeks) from baseline to the end of treatment.
Number of Adverse Events | Every 3 weeks
  Monitoring for safety and toxicity will be performed every cycle (3 weeks) of chemotherapy and whenever patients have problems.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hee Ryu, M.D., Ph.D, Principal Investigator — Asan Medical Center; Young-Iee Park, MD., Ph.D., Principal Investigator — National Cancer Center, Seoul, Korea; Ik-Joo Chung, MD., Ph.D., Principal Investigator — Chonnam National University Hospital
Locations (9):
- South Korea (9):
  - Seoul National University Bundang Hospital, Bundang-gu, Seongnam-si, Gyeonggi-do
  - National Cancer Center, Ilsan, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-eup, Hwasun-gun, Jeollanam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Dongnam Institute of Radiological and Medical Sciences, Busan
  - Yeungnam University Medical Center, Daegu
  - Gangneung Asan Hospital, Gangneung-si
  - Seoul St. Mary's hospital of the Catholic University of Korea, Seoul
  - Asan Medical Center, Seoul

REFERENCES:
- [Background] Ahn YO, Park BJ, Yoo KY, Kim NK, Heo DS, Lee JK, Ahn HS, Kang DH, Kim H, Lee MS, et al. Incidence estimation of stomach cancer among Koreans. J Korean Med Sci. 1991 Mar;6(1):7-14. doi: 10.3346/jkms.1991.6.1.7. PMID 1888453
- [Background] Pyrhonen S, Kuitunen T, Nyandoto P, Kouri M. Randomised comparison of fluorouracil, epidoxorubicin and methotrexate (FEMTX) plus supportive care with supportive care alone in patients with non-resectable gastric cancer. Br J Cancer. 1995 Mar;71(3):587-91. doi: 10.1038/bjc.1995.114. PMID 7533517
- [Background] Glimelius B, Ekstrom K, Hoffman K, Graf W, Sjoden PO, Haglund U, Svensson C, Enander LK, Linne T, Sellstrom H, Heuman R. Randomized comparison between chemotherapy plus best supportive care with best supportive care in advanced gastric cancer. Ann Oncol. 1997 Feb;8(2):163-8. doi: 10.1023/a:1008243606668. PMID 9093725
- [Background] Murad AM, Santiago FF, Petroianu A, Rocha PR, Rodrigues MA, Rausch M. Modified therapy with 5-fluorouracil, doxorubicin, and methotrexate in advanced gastric cancer. Cancer. 1993 Jul 1;72(1):37-41. doi: 10.1002/1097-0142(19930701)72:13.0.co;2-p. PMID 8508427
- [Background] Scheithauer W, Kornek G, Zek B et al. Palliative chemotherapy versus supportive care in patients with metastatic gastric cancer: A randomized trial. Second Int Conf Biol, Prev, Treatm GI Malignancy, Koln, Germany 1995;68(Abstr)
- [Background] Comis RL, Carter SK. A review of chemotherapy in gastric cancer. Cancer. 1974 Nov;34(5):1576-86. doi: 10.1002/1097-0142(197411)34:53.0.co;2-0. No abstract available. PMID 4279136
- [Background] Kaufman S. 5-Fluorouracil in the treatment of gastrointestinal neoplasia. N Engl J Med. 1973 Jan 25;288(4):199-201. doi: 10.1056/NEJM197301252880408. No abstract available. PMID 4264581
- [Background] Schein PS, Macdonald JS, Hoth D, Wooley PV. Mitomycin C: experience in the United States, with emphasis on gastric cancer. Cancer Chemother Pharmacol. 1978;1(2):73-5. doi: 10.1007/BF00254039. No abstract available. PMID 750107
- [Background] Moertel CG, Lavin PT. Phase II-III chemotherapy studies in advanced gastric cancer. Eastern Cooperative Oncology Group. Cancer Treat Rep. 1979 Nov-Dec;63(11-12):1863-9. PMID 393381
- [Background] Lacave AJ, Wils J, Diaz-Rubio E, Clavel M, Planting A, Bleiberg H, Duez N, Dalesio O. cis-Platinum as second-line chemotherapy in advanced gastric adenocarcinoma. A phase II study of the EORTC Gastrointestinal Tract Cancer Cooperative Group. Eur J Cancer Clin Oncol. 1985 Nov;21(11):1321-4. doi: 10.1016/0277-5379(85)90311-6. PMID 4076293
- [Background] Kambe M, Wakui A, Nakao I, Futatsuki K, Sakata Y, Yoshino M, Shimada Y, Taguchi T. A late phase II study of irinotecan (CPT-11) in patients with advanced gastric cancers (abstr 584). Proc Am Soc Clin Oncol 1993;12;198
- [Background] Sulkes A, Smyth J, Sessa C, Dirix LY, Vermorken JB, Kaye S, Wanders J, Franklin H, LeBail N, Verweij J. Docetaxel (Taxotere) in advanced gastric cancer: results of a phase II clinical trial. EORTC Early Clinical Trials Group. Br J Cancer. 1994 Aug;70(2):380-3. doi: 10.1038/bjc.1994.310. PMID 7914428
- [Background] Wagner AD, Grothe W, Haerting J, Kleber G, Grothey A, Fleig WE. Chemotherapy in advanced gastric cancer: a systematic review and meta-analysis based on aggregate data. J Clin Oncol. 2006 Jun 20;24(18):2903-9. doi: 10.1200/JCO.2005.05.0245. PMID 16782930
- [Background] Cunningham D, Starling N, Rao S, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR; Upper Gastrointestinal Clinical Studies Group of the National Cancer Research Institute of the United Kingdom. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008 Jan 3;358(1):36-46. doi: 10.1056/NEJMoa073149. PMID 18172173
- [Background] Kang YK, Kang WK, Shin DB, Chen J, Xiong J, Wang J, Lichinitser M, Guan Z, Khasanov R, Zheng L, Philco-Salas M, Suarez T, Santamaria J, Forster G, McCloud PI. Capecitabine/cisplatin versus 5-fluorouracil/cisplatin as first-line therapy in patients with advanced gastric cancer: a randomised phase III noninferiority trial. Ann Oncol. 2009 Apr;20(4):666-73. doi: 10.1093/annonc/mdn717. Epub 2009 Jan 19. PMID 19153121
- [Background] Koizumi W, Narahara H, Hara T, Takagane A, Akiya T, Takagi M, Miyashita K, Nishizaki T, Kobayashi O, Takiyama W, Toh Y, Nagaie T, Takagi S, Yamamura Y, Yanaoka K, Orita H, Takeuchi M. S-1 plus cisplatin versus S-1 alone for first-line treatment of advanced gastric cancer (SPIRITS trial): a phase III trial. Lancet Oncol. 2008 Mar;9(3):215-21. doi: 10.1016/S1470-2045(08)70035-4. Epub 2008 Feb 20. PMID 18282805
- [Background] Shirasaka T, Shimamato Y, Ohshimo H, Yamaguchi M, Kato T, Yonekura K, Fukushima M. Development of a novel form of an oral 5-fluorouracil derivative (S-1) directed to the potentiation of the tumor selective cytotoxicity of 5-fluorouracil by two biochemical modulators. Anticancer Drugs. 1996 Jul;7(5):548-57. doi: 10.1097/00001813-199607000-00010. PMID 8862723
- [Background] Tatsumi K, Fukushima M, Shirasaka T, Fujii S. Inhibitory effects of pyrimidine, barbituric acid and pyridine derivatives on 5-fluorouracil degradation in rat liver extracts. Jpn J Cancer Res. 1987 Jul;78(7):748-55. PMID 3114201
- [Background] Shirasaka T, Shimamoto Y, Fukushima M. Inhibition by oxonic acid of gastrointestinal toxicity of 5-fluorouracil without loss of its antitumor activity in rats. Cancer Res. 1993 Sep 1;53(17):4004-9. PMID 7689420
- [Background] Yoshisue K, Masuda H, Matsushima E, Ikeda K, Nagayama S, Kawaguchi Y. Tissue distribution and biotransformation of potassium oxonate after oral administration of a novel antitumor agent (drug combination of tegafur, 5-chloro-2,4-dihydroxypyridine, and potassium oxonate) to rats. Drug Metab Dispos. 2000 Oct;28(10):1162-7. PMID 10997934
- [Background] Sakata Y, Ohtsu A, Horikoshi N, Sugimachi K, Mitachi Y, Taguchi T. Late phase II study of novel oral fluoropyrimidine anticancer drug S-1 (1 M tegafur-0.4 M gimestat-1 M otastat potassium) in advanced gastric cancer patients. Eur J Cancer. 1998 Oct;34(11):1715-20. doi: 10.1016/s0959-8049(98)00211-1. PMID 9893658
- [Background] Koizumi W, Kurihara M, Nakano S, Hasegawa K. Phase II study of S-1, a novel oral derivative of 5-fluorouracil, in advanced gastric cancer. For the S-1 Cooperative Gastric Cancer Study Group. Oncology. 2000 Apr;58(3):191-7. doi: 10.1159/000012099. PMID 10765119
- [Background] Fujii M; 0. Chemotherapy for advanced gastric cancer: ongoing phase III study of S-1 alone versus S-1 and docetaxel combination (JACCRO GC03 study). Int J Clin Oncol. 2008 Jun;13(3):201-5. doi: 10.1007/s10147-008-0775-1. Epub 2008 Jun 14. PMID 18553228
- [Background] Jeung HC, Rha SY, Kim HK, Lim HY, Kim S, Kim SY, Gong SJ, Park CH, Ahn JB, Noh SH, Chung HC. Multi-institutional phase II study of S-1 monotherapy in advanced gastric cancer with pharmacokinetic and pharmacogenomic evaluations. Oncologist. 2007 May;12(5):543-54. doi: 10.1634/theoncologist.12-5-543. PMID 17522242
- [Background] Van den Brande J, Schoffski P, Schellens JH, Roth AD, Duffaud F, Weigang-Kohler K, Reinke F, Wanders J, de Boer RF, Vermorken JB, Fumoleau P. EORTC Early Clinical Studies Group early phase II trial of S-1 in patients with advanced or metastatic colorectal cancer. Br J Cancer. 2003 Mar 10;88(5):648-53. doi: 10.1038/sj.bjc.6600781. PMID 12659110
- [Background] Chollet P, Schoffski P, Weigang-Kohler K, Schellens JH, Cure H, Pavlidis N, Grunwald V, De Boer R, Wanders J, Fumoleau P; EORTC Early Clinical Studies Group. Phase II trial with S-1 in chemotherapy-naive patients with gastric cancer. A trial performed by the EORTC Early Clinical Studies Group (ECSG). Eur J Cancer. 2003 Jun;39(9):1264-70. doi: 10.1016/s0959-8049(03)00237-5. PMID 12763215
- [Background] Koizumi W, Tanabe S, Saigenji K, Ohtsu A, Boku N, Nagashima F, Shirao K, Matsumura Y, Gotoh M. Phase I/II study of S-1 combined with cisplatin in patients with advanced gastric cancer. Br J Cancer. 2003 Dec 15;89(12):2207-12. doi: 10.1038/sj.bjc.6601413. PMID 14676796
- [Background] Hyodo I, Nishina T, Moriwaki T, Endo S, Terao T, Hirao K, Nasu J, Hirasaki S, Endo H, Masumoto T, Tajiri H, Kurita A. A phase I study of S-1 combined with weekly cisplatin for metastatic gastric cancer in an outpatient setting. Eur J Cancer. 2003 Nov;39(16):2328-33. doi: 10.1016/s0959-8049(03)00626-9. PMID 14556924
- [Background] Ajani JA, Lee FC, Singh DA, Haller DG, Lenz HJ, Benson AB 3rd, Yanagihara R, Phan AT, Yao JC, Strumberg D. Multicenter phase II trial of S-1 plus cisplatin in patients with untreated advanced gastric or gastroesophageal junction adenocarcinoma. J Clin Oncol. 2006 Feb 1;24(4):663-7. doi: 10.1200/JCO.2005.04.2994. PMID 16446338
- [Background] Lee JL, Kang HJ, Kang YK, Ryu MH, Chang HM, Kim TW, Sohn HJ, Kim H, Lee JS. Phase I/II study of 3-week combination of S-1 and cisplatin chemotherapy for metastatic or recurrent gastric cancer. Cancer Chemother Pharmacol. 2008 Apr;61(5):837-45. doi: 10.1007/s00280-007-0541-5. Epub 2007 Jun 20. PMID 17579864
- [Background] Ohtsu A, Shimada Y, Shirao K, Boku N, Hyodo I, Saito H, Yamamichi N, Miyata Y, Ikeda N, Yamamoto S, Fukuda H, Yoshida S; Japan Clinical Oncology Group Study (JCOG9205). Randomized phase III trial of fluorouracil alone versus fluorouracil plus cisplatin versus uracil and tegafur plus mitomycin in patients with unresectable, advanced gastric cancer: The Japan Clinical Oncology Group Study (JCOG9205). J Clin Oncol. 2003 Jan 1;21(1):54-9. doi: 10.1200/JCO.2003.04.130. PMID 12506170
- [Background] Lee SS, Lee JL, Ryu MH, Chang HM, Kim TW, Kang HJ, Kim WK, Lee JS, Kang YK. Combination chemotherapy with capecitabine (X) and Cisplatin (P) as first line treatment in advanced gastric cancer: experience of 223 patients with prognostic factor analysis. Jpn J Clin Oncol. 2007 Jan;37(1):30-7. doi: 10.1093/jjco/hyl134. PMID 17272321
- [Background] van Meerten E, Eskens FA, van Gameren EC, Doorn L, van der Gaast A. First-line treatment with oxaliplatin and capecitabine in patients with advanced or metastatic oesophageal cancer: a phase II study. Br J Cancer. 2007 May 7;96(9):1348-52. doi: 10.1038/sj.bjc.6603750. Epub 2007 Apr 17. PMID 17437008
- [Background] Louvet C, Andre T, Tigaud JM, Gamelin E, Douillard JY, Brunet R, Francois E, Jacob JH, Levoir D, Taamma A, Rougier P, Cvitkovic E, de Gramont A. Phase II study of oxaliplatin, fluorouracil, and folinic acid in locally advanced or metastatic gastric cancer patients. J Clin Oncol. 2002 Dec 1;20(23):4543-8. doi: 10.1200/JCO.2002.02.021. PMID 12454110
- [Background] Al-Batran SE, Atmaca A, Hegewisch-Becker S, Jaeger D, Hahnfeld S, Rummel MJ, Seipelt G, Rost A, Orth J, Knuth A, Jaeger E. Phase II trial of biweekly infusional fluorouracil, folinic acid, and oxaliplatin in patients with advanced gastric cancer. J Clin Oncol. 2004 Feb 15;22(4):658-63. doi: 10.1200/JCO.2004.07.042. PMID 14966088
- [Background] Lordick F, Lorenzen S, Stollfuss J, Vehling-Kaiser U, Kullmann F, Hentrich M, Zumschlinge R, Dietzfelbinger H, Thoedtmann J, Hennig M, Seroneit T, Bredenkamp R, Duyster J, Peschel C. Phase II study of weekly oxaliplatin plus infusional fluorouracil and folinic acid (FUFOX regimen) as first-line treatment in metastatic gastric cancer. Br J Cancer. 2005 Jul 25;93(2):190-4. doi: 10.1038/sj.bjc.6602697. PMID 16012522
- [Background] Park YH, Kim BS, Ryoo BY, Yang SH. A phase II study of capecitabine plus 3-weekly oxaliplatin as first-line therapy for patients with advanced gastric cancer. Br J Cancer. 2006 Apr 10;94(7):959-63. doi: 10.1038/sj.bjc.6603046. PMID 16552439
- [Background] Neri B, Pantaleo P, Giommoni E, Grifoni R, Paoletti C, Rotella V, Pantalone D, Taddei A, Mercatelli A, Tonelli P. Oxaliplatin, 5-fluorouracil/leucovorin and epirubicin as first-line treatment in advanced gastric carcinoma: a phase II study. Br J Cancer. 2007 Apr 10;96(7):1043-6. doi: 10.1038/sj.bjc.6603644. Epub 2007 Mar 13. PMID 17353926
- [Background] Lee J, Kang WK, Kwon JM, Oh SY, Lee HR, Kim HJ, Park BB, Lim HY, Han MJ, Park JO, Park YS. Phase II trial of irinotecan plus oxaliplatin and 5-fluorouracil/leucovorin in patients with untreated metastatic gastric adenocarcinoma. Ann Oncol. 2007 Jan;18(1):88-92. doi: 10.1093/annonc/mdl317. Epub 2006 Sep 13. PMID 16971670
- [Background] Zhang CX, Huang S, Xu N, Fang JW, Shen P, Bao YH, Mou BH, Shi MG, Zhong XL, Xiong PJ. Phase II study of epirubicin plus oxaliplatin and infusional 5-fluorouracil as first-line combination therapy in patients with metastatic or advanced gastric cancer. Anticancer Drugs. 2007 Jun;18(5):581-6. doi: 10.1097/CAD.0b013e3280146296. PMID 17414627
- [Background] Di Lauro L, Nunziata C, Arena MG, Foggi P, Sperduti I, Lopez M. Irinotecan, docetaxel and oxaliplatin combination in metastatic gastric or gastroesophageal junction adenocarcinoma. Br J Cancer. 2007 Sep 3;97(5):593-7. doi: 10.1038/sj.bjc.6603917. Epub 2007 Jul 31. PMID 17667920
- [Background] Al-Batran SE, Hartmann JT, Probst S, Schmalenberg H, Hollerbach S, Hofheinz R, Rethwisch V, Seipelt G, Homann N, Wilhelm G, Schuch G, Stoehlmacher J, Derigs HG, Hegewisch-Becker S, Grossmann J, Pauligk C, Atmaca A, Bokemeyer C, Knuth A, Jager E; Arbeitsgemeinschaft Internistische Onkologie. Phase III trial in metastatic gastroesophageal adenocarcinoma with fluorouracil, leucovorin plus either oxaliplatin or cisplatin: a study of the Arbeitsgemeinschaft Internistische Onkologie. J Clin Oncol. 2008 Mar 20;26(9):1435-42. doi: 10.1200/JCO.2007.13.9378. PMID 18349393
- [Background] Lee JL, Kang YK, Kang HJ, Lee KH, Zang DY, Ryoo BY, Kim JG, Park SR, Kang WK, Shin DB, Ryu MH, Chang HM, Kim TW, Baek JH, Min YJ. A randomised multicentre phase II trial of capecitabine vs S-1 as first-line treatment in elderly patients with metastatic or recurrent unresectable gastric cancer. Br J Cancer. 2008 Aug 19;99(4):584-90. doi: 10.1038/sj.bjc.6604536. Epub 2008 Jul 29. PMID 18665164
- [Derived] Lee KW, Chung IJ, Ryu MH, Park YI, Nam BH, Oh HS, Lee KH, Han HS, Seo BG, Jo JC, Lee HR, Kim JW, Park SR, Cho SH, Kang YK; SOPP study investigators. Multicenter phase III trial of S-1 and cisplatin versus S-1 and oxaliplatin combination chemotherapy for first-line treatment of advanced gastric cancer (SOPP trial). Gastric Cancer. 2021 Jan;24(1):156-167. doi: 10.1007/s10120-020-01101-4. Epub 2020 Jun 28. PMID 32596783